CLINICAL TRIAL: NCT01431053
Title: Phase 2 Study of Aspirin Plus Exemestane Comparing With Exemestane Alone in the Adjuvant Treatment of Postmenopausal Breast Cancer
Brief Title: Study of Aspirin and Exemestane as Adjuvant Treatment in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Associate Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CH-BC-011
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Breast Neoplasms
Keywords: exemestane; aspirin; quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Aspirin; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exemestane + Aspirin (Experimental)
  Interventions: Drug: aspirin; Drug: Exemestane
- Exemestane (Active Comparator)
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: aspirin — Aspirin 50mg po daily
  Arms: Exemestane + Aspirin
Drug: Exemestane — Exemestane 25mg po daily

SUMMARY:
This is a phase II study to assess efficacy/safety of Exemestane with or without Aspirin as the adjuvant treatment in postmenopausal breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer after surgery postmenopausal

Exclusion Criteria:

* contraindication of aspirin

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China